CLINICAL TRIAL: NCT04599985
Title: Effectiveness of Two Balance Training Protocols on Static and Dynamic Balance, Proprioception, Range of Motion, and Pain in Athletes With Chronic Ankle Instability: A Randomized Comparative Study
Brief Title: Effect of Balance Training Protocols on Balance, Proprioception, ROM, and Pain in Athlete With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-11
Record Dates: First submitted 2020-10-12; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel groups randomized comparative Trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Star excursion balance training (SEBT) (Experimental): Received star excursion balance training (SEBT) program. Performed 3-trials in all 8 directions of the SEBT grid.
  Interventions: Other: star excursion balance training (SEBT)
- Simplified star excursion balance training (SSEBT) (Active Comparator): Received simplified star excursion balance training (SSEBT) program. Performed 3-trials in all 3 directions of SSEBT grid.
  Interventions: Other: Simplified star excursion balance training (SSEBT)

INTERVENTIONS:
Other: star excursion balance training (SEBT) — The SEBT is aimed to be maintained the single limb stance on one leg while reaching farthest possible with the swing leg. An individual can reach farthest with the swing leg while maintaining the balance on the stance leg
  Arms: Star excursion balance training (SEBT)
Other: Simplified star excursion balance training (SSEBT) — It is one of the training protocols, in a simplified way, with respect to star excursion balance test. It consists a series of reaching tasks for the lower limbs in three-directions i.e., anteromedial, medial and posteromedial.
  Arms: Simplified star excursion balance training (SSEBT)

SUMMARY:
The ankle joint sustains injuries particularly in athletics/sports activities at a high rate, resulting in loss of static & dynamic balance, neuromuscular control, and diminished lower extremity's function. This study aimed to compare the effectiveness of two balance-training protocols on balance, proprioception, range of motion (ROM), and pain in male athletes with chronic ankle instability (CAI). Both the balance training protocols were proven to be equally effective in improving the static & dynamic balance, proprioception, ROM, and pain in athletes with CAI.

DETAILED DESCRIPTION:
Injuries to the lower extremity account for 55-90% of all sports injuries. Of these, the knee, ankle, and foot are generally the three most commonly injured anatomic parts in sports. The incidence of ankle injuries is quite high, constituting 20%-25% of all time-loss injuries in every running or jumping sport, including basketball, football, soccer, field hockey, and volleyball. Out of all ankle sprains injuries in sport, 85% cases comprised of lateral ankle sprain (LAS). Up to 74% sufferers of LAS have been accounted for the incidence of chronic ankle instability (CAI). Balance impairments developed as a by-product over extended duration of undermined treatment for ankle injuries. Previous study reported that the dynamic balance greater affected during performing double-leg stance by the patients with CAI than patient with stable ankle when measured by time-to-stabilization (TTS) in the direction of anterior-posterior post tibial nerve stimulation. Thus, concluded that that the value of longer time-to-stabilization indicate an increased relaxation time and after external-perturbation, relatively a longer time needed to identify to a stable pattern.

The management of CAI include both non-surgical and surgical measures. Non-surgical approach includes use of electrical modalities, the rest, ice, compression and elevation of the limb (RICE) principle of therapy for pain relief, functional rehabilitation for gaining strength of the muscles of foot and ankle complex. Moreover, balance training program have been introduced successfully to achieve the static and dynamic balance in order to regain normalcy specially in athletes. Failure of functional rehabilitation indicates for the surgical intervention such as anatomic repair of the anterior talofibular and calcaneofibular ligaments, anatomic reconstruction with autograft or allograft, ankle arthroscopy when intra-articular conditions associated with chronic ankle instability.In literature, there is lack of focus on the Star Excursion Balance Training (SEBT) as well as Simplified Star Excursion Balance Training (SSEBT) which can be used as a balance training protocol for the improvement of dynamic balance especially in the cases of chronic ankle instability. Since, in addition to the static balance, the dynamic balance plays an important role to assesses the balance and neuromuscular control for lower extremity. As lower extremity balance has been linked to the ankle injuries and deteriorated performance in sports.[27]. Hence, the question arises whether a training program using either star excursion balance training (SEBT) or simplified star excursion balance training (SSEBT), can enhance the static and dynamic balance among athletes having chronic ankle instability? A total of 32-participants (male; aged between 18-25 years) with CAI randomly assigned to two groups to receive their postulated balance training protocols. Star excursion balance test, single-leg stance time, foot position sense, visual analog scale, and goniometer were used to assess the dynamic and static balance, proprioception, pain intensity, and ankle ROM respectively at pre-training (baseline) week 1st and post-training week 1st, 2nd, 3rd, and 4th (follow-up).

Both the SEBT and SSEBT protocol proved to be equally effective in the improvement of static & dynamic balance, ankle joint position sense and ROM, and reduction in ankle pain among athletes with CAI. However, SSEBT protocol aid more advantage over SEBT protocol in terms of time consumption and level of muscle fatigue as it consumes less time and produces less fatigue-level because of its (SSEBT) less reaching task (3-directions only) compared to SEBT (8-directions only). Therefore, it is advice to the physical therapist to use the SSEBT protocol while dealing with the problem of static & dynamic balance, joint position sense, ROM, and pain among athletes with CAI.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported case of unilateral CAI with grade I & II verified on CT/MRI by orthopedic surgeon;
* Aged between 18-25 years;
* Onset between 2 to 6 months;
* Exhibited enough strength and flexibility of lower extremity, available ankle ROM, and coordination to execute SEBT and SSEBT.

Exclusion Criteria:

* Self-reported case of bilateral CAI;
* Grade III ankle sprain;
* No past injuries to the lower extremity including ankle sprain within 2-months prior to the commencement of the study;
* Exhibited any neurological, vestibular, and visual disorder;
* Showed muscle tightness, muscle weakness and joint stiffness of lower extremity;
* History of fracture to the ankle; and
* Showed non-cooperation for the study

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Young adult athletes with chronic ankle instability
Enrollment: 32 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Static Balance | 4-weeks
  Static balance assessed by single-leg stance time test with eyes open and closed. It measures the time (in sec) taken by an individual to uphold their base of support with minimal movement while standing on single leg.
Proprioception | 4-weeks
  Assessed by foot position sense. Foot position sense recorded by placing the ankle joint of non-affected side in some degrees of either dorsiflexion or plantarflexion, and asking athlete to match the position with the affected ankle with eyes closed. Angle of difference in the position of ankles was noted in degrees.
Pain intensity, | 4-weeks
  assessed by Visual Analog Scale (VAS). A 10-cm horizontal line marked with 0 (no pain) and 10 (worst pain) on its either end.
Ankle Range of motion | 4-weeks
  Assessed by hand held half-circle goniometer marked with 0 and 180 degree at either end. It has two arm named as stable arm which is fixed in line with the axis of the non-movable arm and movable arm of goniometer is fixed with the movable arm of the body. It is measured in degree.
Dynamic balance | 4-weeks
  The dynamic balance assessed by Star Excursion Balance Test (SEB test) where an individual was asked to stand barefooted on the affected leg and attempt to reach farthest in all 8-directions one by one with the swing leg and return to the starting position while maintaining the balance on the stance leg. Either falling of swing leg or the deviation of stance-leg from its fixed place while attempting to reach farthest in a particular direction and reaching to its starting position considered as a foul to the test and discarded the reading until correct reach performed.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT-Ortho, Principal Investigator — Rehabilitation Research Chair, CAMS, King Saud University, Riyadh, Saudi Arabia
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No